CLINICAL TRIAL: NCT02958345
Title: Placebo Controlled Evaluation of the Cell Mediated Immune Response of Cirrhotic Subjects to Zostavax™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-356128
Record Dates: First submitted 2016-10-24; First posted 2016-11-08 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Herpes Zoster; Fibrosis
MeSH Terms: conditions — Herpes Zoster; Fibrosis | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zostavax (Active Comparator): Subjects will receive 0.65 mL of Zostavax subcutaneously in the deltoid region of the upper arm.
  Interventions: Biological: Zostavax
- Placebo (Placebo Comparator): Subjects randomized to placebo will receive an injection of 0.65 mL of sterile normal saline subcutaneously in the deltoid region of the upper arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Zostavax — Vaccination with one dose of Zostavax per Zostavax package insert
  Other Names: Zoster Vaccine Live
  Arms: Zostavax
Other: Placebo — Injection of 0.65 mL of sterile normal saline
  Arms: Placebo

SUMMARY:
Study Design:

Double-blinded, placebo controlled study of the efficacy of Zostavax in cirrhosis.

Subjects will receive either Zostavax or placebo and will be followed for four months.

Hypothesis:

The investigators hypothesize Zostavax would induce cell-based immunity in cirrhotic patients like that seen in elderly patients.

DETAILED DESCRIPTION:
Study aim, background, and design

Herpes Zoster (Shingles) is a major cause of pain and expense to the elderly and chronically ill. The incidence is estimated at 3 in 1,000 patients. Zostavax™ is a high dose, live varicella vaccine that has been validated in very large placebo control trials to reduce the incidence of Herpes Zoster rash and post herpetic neuralgia in patients over 50 years of age. Additionally the vaccine has been shown to increase quality of life in these patients. Symptomatic Herpes Zoster rates are particularly high post liver transplant with the 3-, 5-, and 10-year actuarial rates of Herpes Zoster of 3%, 10%, 14%, and 18%, respectively. Zostavax is currently recommended for patients prior to solid organ transplantation with no adult data in liver transplant candidates to support that practice. And Although cirrhosis has been acknowledged as a risk factor for symptomatic Herpes Zoster, there is no published data on the efficacy of Zostavax in chronically ill cirrhotic adults pre-transplantation. In particular, it is not known whether or not chronically ill cirrhotic patients demonstrate the appropriate age related cell-mediated immune response seen in the original Zostavax trials.

Procedure

The study will be divided into 3 parts: Screening, Day 1 (or administration of study drug), and Follow Up.

There will be a 4 week screening period. The following procedures will occur in Screening:

Sign consent History and physical exam Inclusion and exclusion review Collection of concomitant medications

The screening visit may occur on the same day as the Day 1 visit. The following procedures will occur on Day 1:

Confirm eligibility Predose lab collection: Interferon-G Enzyme-Linked Immunospot Assay (ELISPOT), GPELISA, VZV Glycoprotein Enzyme-Linked Immunosorbent Assay (also known as Varicella Zoster antibody titre), and Urine pregnancy test for women of childbearing potential Randomize the subject Administer study drug - either Zostavax vaccine or placebo

Follow Up Period:

Month 1 - phone call and collection of adverse events (AEs) and concomitant medications 6 week visit - post dose lab collection: Interferon-G Enzyme-Linked Immunospot Assay (ELISPOT) and GPELISA, VZV Glycoprotein Enzyme-Linked Immunosorbent Assay (also known as Varicella Zoster antibody titre) Months 2, 3 and 4 - phone call and collection of AEs and concomitant medications

Laboratory Tests: The Zoster antibody titer will be run in the Tulane Medical Center Lab and will result in Meditech. The cell mediated immune response lab (ELISPOT) is not a standard lab at Tulane Medical Center. This will be run in Tulane Medical School by a research scientist, whose personal lab has the capabilities to do this special assay.

Telephone Calls: After injection, the subject will follow up with the Investigator as clinically indicated. A study team member will call the subject once a month for 4 months. A standardized approach will be used for every subject. The subject will be asked about concomitant medications and adverse events such as rashes, fevers, hospitalizations, injection site reactions, signs of hepatic decompensation including ascites, confusion, bleeding, and any other physician office visits.

After all of the subjects have completed and assays resulted, the study will be unblinded. The subjects who received placebo will be offered Zostavax vaccine at no cost and will be offered the chance to go into the Follow Up Period described above. The placebo subjects do not have to participate in the Follow Up Period to receive the Zostavax vaccine. The subjects can opt to receive the vaccine or not receive the vaccine or receive the vaccine and give blood on day 1 and again at 6 weeks and also have the option to get the monthly calls for 4 months.

Labs: Pre-vaccination and 6 week post-vaccination measure of varicella immune response Interferon-G Enzyme-Linked Immunospot Assay (ELISPOT) - performed at Tulane Medical School Laboratory.

GPELISA, VZV Glycoprotein Enzyme-Linked Immunosorbent Assay (Varicella Zoster antibody titre) - performed at Tulane Medical Center Laboratory.

There will be approximately 20 cc of blood drawn per lab collection. Total volume of blood drawn for the study is 40cc.

Four month post dose monitoring: telephone contact occurring once a month for 4 months to monitor for adverse events and concomitant medications.

All placebo subjects will be offered complimentary Zostavax vaccine after study closed and un-blinded. See detailed explanation in Procedure.

Randomization:

Thirty subjects will be randomized via sealed envelope system to either vaccine or placebo. Fifteen envelopes will have the Zostavax designation and fifteen envelopes will have the placebo designation. The subject will choose one of the sealed envelopes for treatment. The sealed envelope is taken to the pharmacist who will open the envelope and dispense the treatment as indicated. Only the pharmacist is unblinded to the treatment.

Adverse events:

Adverse Events will be collected from Day 1 until the end of the subject's participation. Events of interest are listed below.

Clinical Herpes Zoster Injection site reaction Hospitalization (any cause) Hepatic decompensation-new onset ascites, encephalopathy, portal hypertensive bleeding or new hepatocellular carcinoma Death

Should the subject have an injury or health problem that is due to taking part in this study, the subject or the subject's insurance will be responsible for the cost. The investigators do not expect any hospitalizations or complications requiring intervention.

Treatment of clinical Herpes Zoster infection:

All subjects who develop a clinical diagnosis of Herpes Zoster during the study will be treated with anti-virals if indicated and appropriate pain relief as needed. The subject or the subject's insurance will be responsible for the cost.

Risks:

There are risks associated with every drug study. The investigators do not suspect that the subjects will be placed at increased risk.

Zostavax: Zostavax is considered very safe, but there are possible side effects, contraindications and warnings/precautions. The following are listed in the Zostavax Package Insert:

Adverse Reactions The most frequent adverse reactions, reported in ≥1% of subjects vaccinated with Zostavax, were headache and injection-site reactions.

Contraindications Hypersensitivity - Zostavax should not be administered to individuals with a history of anaphylactic/anaphylactoid reaction to gelatin, neomycin or any other component of the vaccine.

Immunosuppression - Zostavax is a live, attenuated varicella-zoster vaccine and administration may result in disseminated disease in individuals who are immunosuppressed or immunodeficient. Zostavax should not be administered to immunosuppressed or immunodeficient individuals including those with a history of primary or acquired immunodeficiency states, leukemia, lymphoma or other malignant neoplasms affecting the bone marrow or lymphatic system, AIDS or other clinical manifestations of infection with human immunodeficiency viruses, and those on immunosuppressive therapy.

Pregnancy - Zostavax should not be administered to pregnant women. It is not known whether Zostavax can cause fetal harm when administered to a pregnant woman or can affect reproduction capacity. However, naturally occurring VZV infection is known to sometimes cause fetal harm. Therefore, Zostavax should not be administered to pregnant women, and pregnancy should be avoided for 3 months following administration of Zostavax.

Warnings and Precautions Hypersensitivity Reactions - Serious adverse reactions, including anaphylaxis, have occurred with Zostavax. Adequate treatment provisions, including epinephrine injection (1:1,000), should be available for immediate use should an anaphylactic/anaphylactoid reaction occur.

Transmission of Vaccine Virus - Transmission of vaccine virus may occur between vaccinees and susceptible contacts.

Concurrent Illness - Deferral should be considered in acute illness (for example, in the presence of fever) or in patients with active untreated tuberculosis.

Limitations of Vaccine Effectiveness - Vaccination with Zostavax does not result in protection of all vaccine recipients. The duration of protection beyond 4 years after vaccination with Zostavax is unknown. The need for revaccination has not been defined.

Zostavax is not indicated for nursing mothers. It is unknown if the vaccine is secreted in human milk, therefore, caution should be used in nursing women.

Blood draw: There will be two blood draws 6 weeks apart which should be minimal risk. Risks include bruising, redness, or swelling at the site.

Confidentiality: The identity of all subjects will be protected. Subjects will be assigned a unique identifier. Study related data will be kept in a database under password protection in a locked office. The Key will be stored separately in a locked file cabinet in a locked office. Data will be published and presented with complete anonymity to the subject.

The study team will meet weekly to discuss the trial and evaluate adverse events and unanticipated events. All events will be monitored very closely. The study team will follow injection site reaction, development of Herpes Zoster, hepatic decompensation and any hospitalizations. A thorough history and physical will be done at screening and as needed to reduce the chance of adverse events.

Consent process and documentation

A member of the study team will obtain signed informed consent from each subject participating in the trial after an adequate explanation of the research purpose, personnel, procedures, risks and benefits, and the reiteration that research is voluntary. All of the subject's questions will be answered to his satisfaction. The subject will be given plenty of time to decide on participation and will not be made to feel obligated or coerced.

Obtaining informed consent is a process, not just a document. If the risks change during the course of the project, it may be necessary to re-consent the subjects to ensure they are fully informed and still agree to participate.

The informed consent document will be IRB approved. The signed informed consents will be kept for at least 3 years after the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any etiology diagnosed clinically by labs and imaging or by liver biopsy
* Male or Female age 50 to 70

Exclusion Criteria:

* Active or history of Herpes Zoster
* Anaphylactic allergy to neomycin or gelatin
* Immunosuppressive medication use
* Antiviral medication use
* Known history of HIV
* Known immune deficiency disease
* Active on a liver transplant list
* Known malignancy other than non-melanomatous skin cancer within the past five years.
* History of vaccination with varicella or zoster vaccine
* Pregnant or lactating women
* Prisoners
* Post-transplant patient
* Acute illness

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Balart, MD, Principal Investigator — Tulane University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Background] Schmader KE, Johnson GR, Saddier P, Ciarleglio M, Wang WW, Zhang JH, Chan IS, Yeh SS, Levin MJ, Harbecke RM, Oxman MN; Shingles Prevention Study Group. Effect of a zoster vaccine on herpes zoster-related interference with functional status and health-related quality-of-life measures in older adults. J Am Geriatr Soc. 2010 Sep;58(9):1634-41. doi: 10.1111/j.1532-5415.2010.03021.x. PMID 20863322
- [Background] Herrero JI, Quiroga J, Sangro B, Pardo F, Rotellar F, Alvarez-Cienfuegos J, Prieto J. Herpes zoster after liver transplantation: incidence, risk factors, and complications. Liver Transpl. 2004 Sep;10(9):1140-3. doi: 10.1002/lt.20219. PMID 15350004
- [Background] Danziger-Isakov L, Heeger PS. Clinical utility of measuring T-cell immunity to CMV in transplant recipients. Am J Transplant. 2009 May;9(5):987-8. doi: 10.1111/j.1600-6143.2009.02599.x. No abstract available. PMID 19422327
- [Background] Levin MJ, Oxman MN, Zhang JH, Johnson GR, Stanley H, Hayward AR, Caulfield MJ, Irwin MR, Smith JG, Clair J, Chan IS, Williams H, Harbecke R, Marchese R, Straus SE, Gershon A, Weinberg A; Veterans Affairs Cooperative Studies Program Shingles Prevention Study Investigators. Varicella-zoster virus-specific immune responses in elderly recipients of a herpes zoster vaccine. J Infect Dis. 2008 Mar 15;197(6):825-35. doi: 10.1086/528696. PMID 18419349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zostavax | Placebo
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zostavax | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: ELISPOT, Interferon-G Enzyme-Linked Immunospot Assay
Description: Change in vitro cell-mediated immune response to varicella virus before and after vaccination in subjects receiving Zostavax™ versus those receiving placebo.
Time Frame: Day 1 and 6 weeks
Population: Data was not available for analysis due to laboratory processing error.
Arm/Group | Zostavax | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

2. Secondary Outcome: GPELISA, VZV Glycoprotein Enzyme-Linked Immunosorbent Assay (Aka Varicella Zoster Antibody Titre)
Description: Change in pre and post vaccination Varicella Zoster Virus
Time Frame: Day 1 and 6 weeks
Population: Data was not available for analysis due to laboratory processing error.
Arm/Group | Zostavax | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: Follow-up Period: Month 1, 2, 3, and 4.
Arm/Group | Zostavax | Placebo
All-Cause Mortality (participants affected / at risk) | 1/14 | 2/14
Serious Adverse Events (participants affected / at risk) | 2/14 | 4/14
Other Adverse Events (participants affected / at risk) | 9/14 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zostavax (N=14) | Placebo (N=14)
Death (General disorders) | 1 (1) | 2 (2)
Stroke (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Variceal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased ammonia levels and hyponatremia (General disorders) | 0 (0) | 1 (1)
Decompensated cirrhosis with renal failure (General disorders) | 0 (0) | 1 (1)
Decompensated liver failure (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zostavax (N=14) | Placebo (N=14)
Hyperkalemia (General disorders) | 0 (0) | 1 (1)
Anemia (General disorders) | 0 (0) | 2 (2)
Upper respiratory congestion (Infections and infestations) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Redness at injection site (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Induration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pain at injection site (General disorders) | 2 (2) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Seasonal allergic rhinitis (General disorders) | 1 (1) | 0 (0)
Soreness at injection site (General disorders) | 2 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blocked artery in leg (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Hyperammonemia (General disorders) | 0 (0) | 1 (1)
Acute-on-chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 0 (0) | 1 (1)
Warmth at injection site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Swelling (General disorders) | 2 (2) | 1 (1)
Soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu (Infections and infestations) | 1 (1) | 0 (0)
Bleeding from gums (General disorders) | 1 (1) | 0 (0)
Facial laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomach virus (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Broken rib (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Klebsiella pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No